CLINICAL TRIAL: NCT06706700
Title: Definition of Radiological and Endocrine/metabolic/inflammatory Biomarker(s) to Identify Highgrade Dysplasia/invasive Carcinoma in Patients with Intraductal Papillary Mucinous Neoplasms of the Pancreas
Brief Title: Endocrine, Metabolic, Inflammatory Biomarkers to Identify Highgrade Dysplasia/invasive Carcinoma in Patients with IPMN of the Pancreas
Acronym: EMI-IPMN
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Stefano Crippa, Associate Professor, IRCCS San Raffaele
Other Study IDs: EMI-IPMN
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Intraductal Papillary Mucinous Neoplasm of Pancreas; Pancreatic Cyst
Keywords: ipmn; intraductal papillary mucinous neoplasm of the pancreas; Pancreatic Cysts
MeSH Terms: conditions — Pancreatic Intraductal Neoplasms; Pancreatic Cyst

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples from peripheral and portal blood: Serum, Plasma, PBMCs and whole blood will be stored; Cyst Fluid from the pancreatic cyst; Formalin-Fixed Paraffin-Embedded tissue from the Pancreatic Cyst
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort A: A retrospective study of a cohort of 350 resected patients with a histologically-confirmed IPMN, diagnosed from the 1st January 2009 to the 31st May 2018 following these inclusion criteria:
  * histologically proven IPMNs with full pathological data (type of IPMNs, grade of dysplasia; for invasive IPMNs: grading, pTNM classification, presence of perineural (microvascular infiltration)
  * availability of clinical and imaging criteria for surgical resections defined by International and European guidelines (worrisome features and high-risk stigmata according to International Guidelines and absolute/relative criteria for surgery according to European guidelines
  * age ≥18 years and exclusion criteria:
  * lack of preoperative clinical and radiological data according the two guidelines
- Cohort B: A prospective observational study whose aim is to identify EMI profiles and radiological/endosonographical biomarker(s) associated to surgically removed IPMNs with HGD/IC.
  Patients diagnosed with IPMN and candidates for resection with following inclusion criteria will be enrolled:
  * Age >= 18 years
  * Charlson comorbidity index <7 [26] The patients' cohort will be selected following the best criteria for surgery identified in the retrospective study (Cohort A).
  At the admission, patients will be informed by PI, or his delegates about the study, and they will be asked to sign the specific informed consents (see par. 5.1) In the course of standard pre-operative evaluation, all patients will undergo MRI and EUS, within no more than 3 months between exams.
- Cohort C: A prospective study with the aim to validate potential biomarker(s) identified in the Cohort B.
  Patients with a diagnosis of IPMN candidate for resection with the following inclusion criteria will be enrolled:
  * Age >= 18 years
  * Charlson comorbidity index <7 [26] The patients' cohort will be selected following the best criteria for surgery identified in the retrospective study (Cohort A).
  At the admission patients will be informed by PI or his delegates about the study and they will be asked to sign specific informed consents

SUMMARY:
Under the hypotheses that a more accurate patients selection could limit the problem of overtreatment and that benign intraductal papillary mucinous neoplasms (IPMN) have a distinguishable Endocrine/Metabolic/Inflammatory (EMI) profile from those with high-grade disease/invasive carcinoma, this study has three specific aims. The first aim is to evaluate and confirm the accuracy of the updated versions of International and European guidelines for the management of IPMN and it will be addressed by retrospectively applying the criteria included in the two guidelines on 350 patients with resected IPMN in order to determine the most accurate criteria to identify High Grade Dysplasia(HGD)/Invasive Carcinoma (IC).

The second aim is to identify pre-operative biological and/or radiological/endosonographic biomarker(s) able to distinguish low- versus high-risk IPMN for cancer progression in a prospective study by enrolling a cohort of 186 (of which 145 surgically-resected) patients.

The third aim is to prospectively validate biological and/or radiological/endosonographic biomarker(s) (previously identified and optimized) on a new cohort of 50 patients with IPMN undergoing surgical resection.

DETAILED DESCRIPTION:
Up to 40% of patients (pts) undergoing abdominal imaging harbor unsuspected pancreatic cysts, the majority of which intraductal papillary mucinous neoplasms (IPMN). IPMNs are well-known precursors of pancreatic ductal adenocarcinoma (PDAC) without an established temporal window of progression. Current guidelines identify high-risk stigmata (HRS)/absolute criteria(AC) and worrisome features(WF)/relative criteria(RC) as indications for surgical resection of IPMN. Previous guideline criteria were found to be associated with high sensitivity but low specificity for malignancy, resulting in an overtreatment of benign IPMNs, a clinical relevant issue considering the high morbidity/mortality of pancreatectomy. Currently, there are no available hematic biomarkers in peripheral blood, be they DNA, RNA or protein-based, which can identify High Grade Dysplasia(HGD)/Invasive Carcinoma (IC). DNA-based molecular testing of pancreatic cyst fluid obtained during endoscopic ultrasound (EUS)/surgery have been developed and are used to identify advanced neoplasia, with good sensitivity/specificity, and therefore hypothetically, an IPMN HGD/IC-based biomarker could be more readily detected in cyst fluid or in portal blood. This strategy, however has a number of limitations: i) it is highly invasive and costly ii) poor quantity and quality of cyst fluid may lead to incorrect detection (false negatives in molecular testing) ; and iii) a lack of predictive potential of progression over time. New diagnostic tools based on samples of portal blood obtained during EUS or potentially peripheral samples (of new biomarkers) may overcome these limitations.

PDAC has been associated with altered inflammatory and endocrine/metabolic profiles but limited data are available on IPMN and other precursors. Inflammation and malignant progression have become cardinal in cancer research. Tumor-associated neutrophils and cytokines, including TNFalpha and IL-1ß, have been associated with malignant progression also in IPMN. About 40-70% of patients with PDAC experience diabetes or alterations of glucose homeostasis. Diabetes-induced hyperglycemia, hyperinsulinemia, altered insulin-like growth factors production, chronic inflammation and metabolic syndrome have been associated with cancer . In a large cohort of resected IPMNs, preoperative diabetes was significantly associated with HGD/IC, and the risk of IC was highest in patients with recent-onset diabetes.

Obesity is also a well-known risk factor for PDAC; proinflammatory cytokines, known as adipokines are released mainly from visceral adipose tissue stimulating aberrant angiogenesis. An association between visceral obesity and pancreatic fatty infiltration with poor survival was found in PDAC patients. In the setting of IPMN, in a very small cohort of resected patients, significantly higher BMI was associated to an increased rate of malignant IPMN.

EUS, Computed tomography(CT) and magnetic resonance imaging(MRI) are of use in current clinical practice to study and monitor pancreatic diseases. They are all imaging techniques that allow to characterize pancreatic alterations and simultaneously detect endocrino-metabolic alterations (i.e.visceral obesity, liver steatosis, pancreatic fatty infiltration) that may be associated to pancreatic diseases.

Current literature is still debating the superiority of radiological imaging (specifically MRI) or endoscopic ultrasound in identifying worrisome features/high risk stigmata and in correctly distinguishing benign/malignant IPMNs. Preliminary analysis performed in the context of this study, specifically in retrospective Cohort A, aimed at validating International and European guidelines, supports an important role for EUS in identifying risk of malignancy in IPMNs. In fact, 31/116 patients (26.7%) with WF at MRI were "upstaged" by EUS and the majority of these (77.4%) had malignancy at final pathology. Furthermore, EUS confirmed MRI findings in 87.5% of cases, including 72.4% of radiological WF.

The association among obesity, diabetes, inflammation, alterations of specific endocrine/metabolic pathways and pancreatic cancer development from its precursors (IPMN) are more complex, and needs further investigations.

The driving hypotheses of this study are that i) a more accurate patients selection could limit the problem of overtreatment, ii) that benign/indolent IPMN have a distinguishable Endocrine/Metabolic/Inflammatory (EMI) profile from those with HGD/IC, and therefore this research has the following three specific aims.

Aim 1: To retrospectively evaluate and to validate the updated versions of International and European guidelines for the management of IPMN (Cohort A) Aim 2: To identify pre-operative biological and/or imaging biomarker(s) to distinguish low- versus high-risk IPMN for cancer progression in a prospective study of surgically-resected patients (Cohort B) Aim 2.1: To compare MRI and EUS in the pre-operative evaluation of IPMNs and with respect to pathological findings. In particular, primary endpoint will be the identification of main pancreatic duct involvement. Secondary endpoints will be evaluation of the degree of main duct involvement (extension of IPMN involvement, MPD diameter at predetermined points, maximum diameter of MPD), the presence of thickened ductal walls, mural nodules and the characteristics of the surrounding parenchyma (fatty infiltration/vanishing pancreas).

Aim 3: To prospectively validate biological and/or imaging biomarker(s) previously identified (Aim 2) on patients with IPMN undergoing surgical resection (Cohort C)

ELIGIBILITY:
cohort A: inclusion criteria:

* histologically proven IPMNs with full pathological data (type of IPMNs, grade of dysplasia; for invasive IPMNs: grading, pTNM classification, presence of perineural (microvascular infiltration)
* availability of clinical and imaging criteria for surgical resections defined by International and European guidelines (worrisome features and high-risk stigmata according to International Guidelines and absolute/relative criteria for surgery according to European guidelines
* age ≥18 years

exclusion criteria:

- lack of preoperative clinical and radiological data according the two guidelines

Cohort B and C:

inclusion criteria:

* Age >= 18 years
* Charlson comorbidity index <7
* indication for surgery for suspected IPMN

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be enrolled in the outpatient clinic, if they meet the required criteria for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 586 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
evaluation of the best guideline between the International and European guidelines | from the collection of the retrospective cohort to 12 months
  The criteria included in the two guidelines will be retrospectively applied on 350 patients with resected IPMN. Clinical pathological and imaging data will be retrieved from institutional archives systems.
  As we may be not able to identify a more accurate guideline, we may select specific criteria from each of the two guidelines, thus selecting p batients for surgery based on a combination of criteria from both guidelines.
  The identified best criteria will be applied to select the discovery cohort and the validation cohort of the prospective studies.
endocrine, metabolic and inflammatory profile | from the enrollment to 8 month
  The following parameters will be measured in peripheral and portal serum/plasma and in the cyst fluid with commercially available kits
imaging-based biomarker(s) | at the time of enrollment
  As per standard-of-care current clinical practice in our institution, all patients will undergo 1.5T contrast-enhanced MR cholangiopancreatography (MRCP) with 3D acquisition protocol of the pancreatic ducts/ biliary tree
evaluation of the accuracy of the biomarkers in predicting the pathological diagnosis | at the end of the enrollment
  the accuracy at identifying malignant IPMN of the identified biomarkers will be tested.

SECONDARY OUTCOMES:
evaluation of the accuracy of the MRI versus the EUSP in identifying the involvement of the main pancreatic duct | at the end of the enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes